CLINICAL TRIAL: NCT05790902
Title: COMPARISON OF SILODOSIN AND TAMSULOSIN IN MEDICAL EXPULSIVE THERAPY OF DISTAL URETERIC CALCULI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, AJ Arif, DR ABDUL JABBAR ARIF, Armed Forces Institute of Urology, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFIU-2022-02
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Silodosin, Tamsulosin, Medical Expulsive Therapy, Distal Ureteric Calculi
MeSH Terms: interventions — silodosin; Tamsulosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silodosin Group (Experimental): The patients used Silodosin for ureteric calculi
  Interventions: Drug: Silodosin
- Tamsulosin Group (Experimental): The patients used Tamsulosin for ureteric calculi
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Silodosin — The patients used Silodosin for Medical expulsive therapy of ureteric calculi
  Arms: Silodosin Group
Drug: Tamsulosin — The patients used Tamsulosin for Medical expulsive therapy of ureteric calculi
  Arms: Tamsulosin Group

SUMMARY:
to compare efficacy and safety of Silodosin and Tamsulosin in Medical expulsive therapy of Distal Ureteric Calculi.

DETAILED DESCRIPTION:
to compare efficacy and safety of Silodosin and Tamsulosin in Medical expulsive therapy of Distal Ureteric Calculi in our local setup to find out the optimal drug which promptly and quickly cures the disease thus enabling the person to return to routine activity with less adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic, unilateral, single, uncomplicated Distal Ureteric Calculi of <10 mm in size (on plain CT KUB)

Exclusion Criteria:

* solitary kidney, bilateral ureteric stones, UTI, renal impairment, high-grade hydronephrosis (Grades 3 and 4), any history of previous endoscopic or surgical interventions, pregnancy, diabetes mellitus,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Stone clearance rate | upto 4 weeks
  Stone clearance rate

SECONDARY OUTCOMES:
Stone expulsion time | upto 4 weeks
  Stone expulsion time

CONTACTS AND LOCATIONS:
Locations (1):
- AFIU Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No